CLINICAL TRIAL: NCT05303584
Title: Immunogenicity and Safety of the Heterologous Prime-boost Immunization with an Adenovirus Type-5 Vector-based COVID-19 Vaccine (Ad5-nCoV) After Three-dose Priming with an Inactivated COVID-19 Vaccine in Adults Aged 18 Years and Above: a Randomized, Open-label, Parallel-controlled Clinical Trial
Brief Title: Heterologous Boost Immunization with Ad5-nCoV After Three-dose Priming with an Inactivated SARS-CoV-2 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT153
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Ad5-nCoV; Inactivated Vaccine; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Approximately 70 subjects recruited from the prior clinical trial and newly enrolled 50 subjects will receive a booster dose of aerosolized Ad5-nCoV after three-dose priming with ICV
  Interventions: Biological: Ad5-nCoV-IH
- Group B (Experimental): Approximately 70 subjects recruited from the prior clinical trial and newly enrolled 50 subjects will receive a booster dose of intramuscular Ad5-nCoV after three-dose priming with CoronaVac
  Interventions: Biological: Ad5-nCoV-IM
- Group C (Experimental): Approximately 70 subjects recruited from the prior clinical trial and newly enrolled 50 subjects will receive homologous fourth dose of CoronaVac.
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: Ad5-nCoV-IH — The orally aerosolized Ad5-nCoV is a replication defective Ad5 vectored COVID-19 vaccine expressing the full-length spike gene of wide-type SARS-CoV-2, Wuhan-Hu-1. The Ad5-nCoV vaccine was supplied in 1.5mL/vial, at a concentration of 1.0 × 1011 viral particles per mL as a liquid formulation. 0.1 ml of Ad5-nCoV vaccine will be aerosolized by using Continuous Vapouring System. Then, the aerosolized droplets will be poured into a disposable suction cup and be inhaled by participants through mouth.
  Other Names: aerosolized Ad5-nCoV; Convidecia
  Arms: Group A
Biological: Ad5-nCoV-IM — The Ad5-nCoV is a replication defective Ad5 vectored COVID-19 vaccine expressing the full-length spike gene of wide-type SARS-CoV-2, Wuhan-Hu-1. It was supplied in 1·5mL/vial, at a concentration of 1.0 × 1011 viral particles per mL as a liquid formulation. Participants will be administrated 0.5ml（5×1010VP）of Ad5-nCoV vaccine intramuscularly.
  Other Names: intramuscular Ad5-nCoV
  Arms: Group B
Biological: CoronaVac — CoronaVac is an inactivated whole-virion vaccine with aluminium hydroxide as the adjuvant, prepared with a novel coronavirus (CZ02 strain) inoculated in African green monkey kidney cells (Vero cells). One dose of CoronaVac contains 3 μg of SARS-CoV-2 virion in a 0.5 mL aqueous suspension for injection with 0.45 mg/mL of aluminium.
  Arms: Group C

SUMMARY:
This is an open-label, randomized, parallel-controlled clinical trial to evaluate the safety and immunogenicity of heterologous prime-boost immunization with an aerosolized (Ad5-nCoV-IH) or intramuscular (Ad5-nCoV-IM) Ad5-nCoV after three-dose priming with an inactivated COVID-19 vaccine (CoronaVac) in adults aged 18 years and above. A total of 360 subjects will be included. Approximately 210 subjects who have completed three doses of CoronaVac more than 6 months ago in the prior clinical trial and other 150 eligible subjects will be recruited and randomized respectively in a ratio of 1:1:1 to receive a booster dose of Ad5-nCoV-IH or Ad5-nCoV-IM or ICV. The occurrence of adverse reactions within 28 days and serious adverse events within 6 months after vaccination will be observed in all participants. In addition, blood and saliva samples will be collected from all participants on the day 0 before and 14, 28 days and 3, 6 months after the booster vaccination. Each subject will remain in this study for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Health subjects aged ≥18 years
* The subject can provide with informed consent and sign informed consent form (ICF).
* The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the 6-month follow-up of the study.
* Participants who have received three-dose of inactivated SARS-CoV-2 vaccine more than 6 months ago.

Exclusion Criteria:

* Have the medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* Be allergic to any component of the research vaccines, or used to have a history of hypersensitivity or serious reactions to vaccination.
* Vaccine-related SAE occurred after previous vaccination with COVID-19 vaccine.
* Women with positive urine pregnancy test or in lactation.
* Have acute febrile diseases or infectious diseases or have a history of SARS.
* Axillary temperature>37.0℃
* Have serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension that cannot be controlled by medication (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg when measured in the field)
* Have severe chronic diseases or condition is not stable, such as asthma, diabetes, thyroid disease
* Congenital or acquired angioedema / neuroedema.
* Have the history of urticaria 1 year before.
* Have asplenia or functional asplenia.
* Patients with chronic obstructive pulmonary disease, pulmonary fibrosis and other pulmonary abnormalities.
* Have history of SARS-CoV-2 infection or COVID-19.
* Have symptoms of upper respiratory tract infection.
* Have traveled to medium or high risk areas or traveled abroad in the past 21 days, and epidemiologically contacted with SARS-CoV-2.
* Any medical, psychological, social, or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2022-04-23 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions within 28 days after the booster dose | Within 28 days the booster dose
  Incidence of adverse reactions within 28 days after the booster dose.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose. | On day 28 after the booster dose
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose.

SECONDARY OUTCOMES:
Geometric Mean Fold Increase (GMI) and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose. | On day 28 after the boost vaccination
  GMI and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose in immunogenicity cohort.
GMT, GMI and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 14, month 3 and 6 after the booster dose. | On day 14, month 3 and 6 after the booster dose
  GMT, GMI and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus as compared to baseline on day 14, month 3 and 6 after the booster dose.
Geometric mean concentration (GMC), GMI and seroconversion of anti-SARS-CoV-2 NP-specific, RBD-specific and NTD-specific IgG measured by ELISA on day 14, day 28 and month 3 and 6 after the booster dose. | On day 14, day 28 and month 3 and 6 after the booster dose
  Geometric mean concentration (GMC), GMI and seroconversion of anti-SARS-CoV-2 NP-specific, RBD-specific and NTD-specific IgG measured by ELISA on day 14, day 28 and month 3 and 6 after the booster dose.
Incidence of adverse reactions within 30 minutes after the booster dose. | Within 30 minutes after the booster dose
  Incidence of adverse reactions within 30 minutes after the booster dose.
Incidence of adverse reactions within 14 days after the booster dose. | Within 14 days after the booster dose
  Incidence of adverse reactions within 14 days after the booster dose.
Incidence of adverse events within 28 days after the booster dose. | Within 28 days after the booster dose
  Incidence of adverse events within 28 days after the booster dose.
Incidence of serious adverse events (SAE) until 6 months after the booster dose. | Within 6 months after the booster dose
  Incidence of SAE until 6 months after booster vaccination.

OTHER OUTCOMES:
GMT, GMI and seroconversion of neutralizing antibodies against VOC/VOI of SARS-CoV-2 virus on day 28 after the booster dose. | On day 28 after the booster dose
  GMT, GMI and seroconversion of neutralizing antibodies against VOC/VOI of SARS-CoV-2 virus on day 28 after the booster dose.
The levels of IFN-γ、TNF-α、IL-2 secreted by specific T cells stimulated with a peptide pool covering the full-length spike glycoprotein on day 14 after the booster vaccination. | On day 14 after the booster vaccination
  The levels of IFN-γ、TNF-α、IL-2 secreted by specific T cells stimulated with a peptide pool covering the full-length spike glycoprotein on day 14 after the booster vaccination.
The levels of anti-SARS-CoV-2 RBD-specific binding IgA in saliva on day 14, day 28 and month 3 and 6 after the booster dose. | On day 28 after the booster dose
  The levels of anti-SARS-CoV-2 RBD-specific binding IgA in saliva on day 14, day 28 and month 3 and 6 after the booster dose.
GMT and GMI of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose stratified by age (aged 18-59 years and over 60 years). | On day 28 after the booster dose
  GMT and GMI of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose stratified by age (aged 18-59 years and over 60 years).
The levels of anti-SARS-CoV-2 N protein binding IgG on day 14 after the booster dose. | On day 14 after the booster dose
  The levels of anti-SARS-CoV-2 N protein binding IgG on day 14 after the booster dose.
The GMT of neutralizing antibodies against the Ad5 before vaccination and any exploratory analyses of other indicators stratified by pre-existing anti-Ad5 NAb titres at baseline（>1:200，≤1:200） | On day 0 before the booster dose
  The GMT of neutralizing antibodies against the Ad5 before vaccination and any exploratory analyses of other indicators stratified by pre-existing anti-Ad5 NAb titres at baseline（>1:200，≤1:200）

CONTACTS AND LOCATIONS:
Overall Officials: Jingxin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia X, Tan ZM, Wan P, Zheng H, Tang R, Chen XQ, Guo XL, Zhu T, Feng JL, Zhong J, Li XL, Zhang ZY, Zhu FC, Li JX. Environmental Impact Assessment for the Use of an Orally Aerosolized Adenovirus Type-5 Vector-Based COVID-19 Vaccine in Randomized Clinical Trials. J Infect Dis. 2023 Sep 15;228(6):715-722. doi: 10.1093/infdis/jiad134. PMID 37202147
- [Derived] Tang R, Zheng H, Wang BS, Gou JB, Guo XL, Chen XQ, Chen Y, Wu SP, Zhong J, Pan HX, Zhu JH, Xu XY, Shi FJ, Li ZP, Liu JX, Zhang XY, Cui LB, Song ZZ, Hou LH, Zhu FC, Li JX; CanSino COVID-19 Study Group. Safety and immunogenicity of aerosolised Ad5-nCoV, intramuscular Ad5-nCoV, or inactivated COVID-19 vaccine CoronaVac given as the second booster following three doses of CoronaVac: a multicentre, open-label, phase 4, randomised trial. Lancet Respir Med. 2023 Jul;11(7):613-623. doi: 10.1016/S2213-2600(23)00049-8. Epub 2023 Mar 7. PMID 36898400